CLINICAL TRIAL: NCT06349096
Title: Open-Label, Safety And Efficacy Investigation Of The Effects Of ClearLift Q-Switched Nd:Yag 1064nm Laser Module In The Treatment Of Facial Skin Wrinkles
Brief Title: Safety And Efficacy Investigation Of The Effects Of ClearLift Q-Switched Nd:Yag 1064nm Laser Module In The Treatment Of Facial Skin Wrinkles
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alma Lasers (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALM-HAR-CLL-23-01
Record Dates: First submitted 2024-03-21; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Facial Skin Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser treatment (Experimental): Treatment of facial skin wrinkles using the Alma Harmony platform with the ClearLift high power Q-switched (QS) 1064nm Nd:YAG laser module
  Interventions: Device: Alma Harmony

INTERVENTIONS:
Device: Alma Harmony — The ClearLift is a class IIb medical device, High Power Q-switched (QS) 1064nm Nd:YAG laser module in the Harmony system. It has a targeted laser module for the non-invasive removal of various colored tattoos, as well as deep and superficial benign pigmented lesions, wrinkles, fine lines, and skin tightening.
  Other Names: ClearLift applicator

SUMMARY:
Alma Lasers ClearLift is a fractional non-ablative Q-Switched laser, allowing practitioners to use the benefits of a high intensity QS laser for the treatment of aged skin. Alma Harmony ClearLift uses a fractional QS laser to achieve a deep mechanical effect beneath the epidermis via a photoacustic effect. This creates a controlled dermal wound while leaving the epidermis intact. The wound healing process stimulates growth of new collagen, skin contracture and tightening. This procedure is virtually painless with no downtime and is safe for all skin types.

Based on this background, we have considered an interest to design a study aimed at assessing the efficacy and safety of a treatment course with ClearLift Module in patients with facial skin wrinkles

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged ≥ 35 and ≤ 55 years
* Presence of type 1-3 facial skin wrinkles, according to the Glogau scale;
* Subjects in reasonably good general health, according to Investigator's judgment;
* Subjects who agree to avoid tanning during the entire investigational period;
* Subjects who agree to avoid any other facial procedure during the entire investigational period; including but not limited to: injectables or threads, peeling of any kind, dermabrasion, facial hair removal or application of any cosmoceutical/pharmaceutical without the consent from the PI only.
* Subjects able to understand the full nature and the purpose of the investigation, including possible risks and side effects, able to cooperate with the Investigator and to comply with the requirements of the entire investigation (ability to attend all the planned investigation visits according to the time limits included) based on Investigator's judgement.
* Subjects willing to sign an informed consent, consent to use their photos for future scientific or marketing purposes, according to the sponsor's needs.

Exclusion Criteria:

* Subjects with active infections;
* Subjects with history of keloid scarring or hypertrophic scar formation;
* Subjects with previous medical treatment of the area, or oral retinoid drug prescribed within the past six months;
* Subjects who have been tanning within the past 30 days;
* Previous surgical treatment of the area selected for the treatment with the investigational device;
* Subjects with any inflammatory skin condition e.g., eczema, active herpes simplex, etc. at the treatment site;
* Subjects with presence of tattoos at the treatment site;
* Subjects with skin cancer or any other cancer and/or any cancer drug therapy (such as ducabaxine, fluorouracil, methotrexate, etc.);
* Subjects with history of autoimmune disorder or evidence of immunosuppression;
* Subjects with cellulitis;
* Subjects with collagen vascular diseases;
* Subjects with thrombocytopenia;
* Subjects with peripheral vascular disease;
* Subjects with Melasma;
* Pregnant or lactating subjects.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-03-26 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | at the 3-month follow-up
  70% of participants will demonstrate any improvement in the treated facial skin wrinkles after ClearLift treatment based on the rating of three blinded assessors that will compare the baseline 2D photographs with the 3-month follow-up visit photographs and will rate the degree of improvement using the 5-points Global Aesthetic Improvement Scale (GAIS)- in which 1 denotes "Wors";2 denotes "No change";3 denotes "Improved"; 4 denotes "Much improved"; and 5 denotes "Very much improved".

SECONDARY OUTCOMES:
Secondary endpoint | at the 1-month follow-up
  Improvement in the treated facial skin wrinkles after ClearLift treatment based on the rating of the investigator that will compare the baseline 2D photographs with the 1-month follow-up visit photographs and will rate the degree of improvement using the 5-points Global Aesthetic Improvement Scale (GAIS)- in which 1 denotes "Wors";2 denotes "No change";3 denotes "Improved"; 4 denotes "Much improved"; and 5 denotes "Very much improved".
Secondary endpoint | at the 1 and 3-month follow-up
  Improvement in skin texture of the treated facial skin wrinkles, as evaluated by the VISIA 3D camera, at the 1- and 3-month follow-up visits compared to baseline
Secondary endpoint | at the 1 and 3-month follow-up
  Participant's satisfaction with treatment at the 1- and 3-month follow-up visits, as evaluated using a 5-point Likert scale, in which 1 denotes "Very dissatisfied";2 denotes "Dissatisfied";3 denotes "Satisfied"; 4 denotes "Very satisfied"; and 5 denotes "Extremely satisfied ".

OTHER OUTCOMES:
Safety & Tolerability | throughout the study
  At the beginning of each visit starting the second treatment visit, the investigator will record the occurrence of adverse events (such as prolonged Erythema/ Edema, Burns, Hematoma / Ecchymosis, Scarring, and Hyperpigmentation.) and will rate their severity according to a 3 points scale in which 1= mild; 2= moderate, and 3=severe.
Safety & Tolerability | immediately after each treatment session (up to 1 month)
  Pain level using a 11- points Numerical Pain Rating Scale (NPRS) in which 0= "No pain" and 10="Worst possible pain", as evaluated at each treatment visit at the end of each treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Arminda Avdulaj, MD, Principal Investigator — Head of San Luca Medical Clinic, Tirana, Albania
Locations (1):
- San Luca Medical Clinic, Tirana, Albania